CLINICAL TRIAL: NCT03503461
Title: Evaluation of the Prevalence of an Hyperactivation of NCC Cotransporter Three Months After Kidney Transplantation in Recipients Treated by Calcineurin Inhibitors
Brief Title: Major Activation Of NCC in Graft Urinary Exosomes
Acronym: MANGUE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/08
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Kidney Transplantation
Keywords: Calcineurin inhibitors; hypertension; kidney transplant; acidosis; Gordon syndrome
MeSH Terms: conditions — Hypertension; Acidosis; Gordon syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Control group is a population of subjects admitted to day hospitalization for renal function tests or in conventional hospitalization, but without kidney transplant. Exosome analysis will be perform in urine sample.
  Interventions: Other: exosomes analysis
- Kidney transplants group: Kidney transplants group is a kidney transplant subjects population 3 months ago. Exosome analysis will be perform in urine sample collected at 3 months.
  Interventions: Other: exosomes analysis

INTERVENTIONS:
Other: exosomes analysis — Perform exosomes analysis in urine sample obtain from usual urine testing in both kidney transplant and control group.

SUMMARY:
Hypertension is common disorder after renal transplantation and is associated with mortality. Calcineurin Inhibitor (CNI), by activating NCC cotransporter, may be a major determinant of hypertension, included in a "Gordon like" syndrome. However, prevalence of NCC activation by CNI is unknown. Our objective is to determine the prevalence of NCC activation three months after transplantation in patient treated by CNI.

DETAILED DESCRIPTION:
Hypertension is common disorder after renal transplantation and is associated with mortality. Calcineurin Inhibitor (CNI), by activating NCC cotransporter, may be a major determinant of hypertension, included in a "Gordon like" syndrome. Gordon syndrome is a rare genetic disorder where NCC cotransporter is overactivated and cause hypertension, metabolic acidosis and tendency to hyperkaliemia. Few studies evaluated NCC expression by exosomes techniques in human kidney transplant, and mostly compared NCC expression in specific subpopulation (for example with or without hypertension). Thus, prevalence of NCC activation by CNI is unknown. To determine it, we will include prospective patients in Bordeaux and la Réunion who undergo urine and blood tests three months after transplantation, and a control group with no transplantation and no use of CNI. First, we will compare kidney recipients and control and use immunoblot to quantify NCC expression in urinary exosomes to identify the population of transplanted with a high activation. Then, we will analyze the relationship between NCC activation and clinicobiological features of Gordon's syndrome.

ELIGIBILITY:
For kidney transplant group :

* inclusion criteria:

  * Age≥18years
  * Recipients three months after kidney transplantation using calcineurin inhibitors
  * Glomerular Filtration Rate>15ml.mn.m2 CKD-EPI
  * Renal ultrasound underwent before inclusion
  * No opposition at participating at the research
* exclusion criteria:

  * Use of diuretic thiazides or aldosterone receptor antagonists in the month preceding inclusion
  * Graft artery stenosis with indication of interventional radiology or surgery

For control group :

* Inclusion criteria

  * No previous transplantation
  * Age≥18years
  * No hypertension
  * No metabolic disorders (dysnatremia, dyskaliemia, acidosis or alkalosis)
  * No opposition at participating at the research
* Exclusion criteria:

  * Use of diuretic thiazides or aldosterone receptor antagonists in the month preceding inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Kidney transplant group is a population of transplant subjects treated with anticalcineurin since 3 months.
  Control group is a population of subjects admitted to day hospitalization for renal function tests or in conventional hospitalization, but without kidney transplant.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
NCC cotransporter expression | Inclusion day
  Dosage of NCC cotransporter expression in urinary exosomes samples in both groups.

SECONDARY OUTCOMES:
Phosphorylated NCC cotransporter expression | Inclusion day
  Dosage of phosphorylated NCC cotransporter expression in urinary exosomes samples in both groups.
pendrine expression in kidney transplant group | Inclusion day
  Dosage of pendrine expression in urinary exosomes samples in kidney transplant group.

CONTACTS AND LOCATIONS:
Locations (2):
- Hopital Pellegrin - Service Néphrologie, transplantation, dialyse et aphérèse, Bordeaux, France
- Hopital Felix Guyon - Service d'Explorations Fonctionnelles Rénales, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No